CLINICAL TRIAL: NCT03924570
Title: Multicenter Study to Reduce Adverse Events in Pediatric Intensive Care Units in Argentina Using a Program to Improve the Transfer of Patients
Brief Title: Reducing Adverse Events in Pediatric Intensive Care Units in Argentina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Hospital JP Garrahan (Other Government); Ministry of Public Health, Argentina (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NRU3126
Record Dates: First submitted 2018-12-12; First posted 2019-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Medical Errors; Preventable Adverse Events

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive training in the use of the IPASS package to improve communications during hands off.
  Interventions: Behavioral: IPASS
- Control (No Intervention): Until randomization this arm will continue running hands offs per usual care.

INTERVENTIONS:
Behavioral: IPASS — IPASS is behavioral package to improve transitions of care by providing a framework to hands off.
  Arms: Intervention

SUMMARY:
Introduction: Errors in communication, and during transfers of information and medical responsibility, are frequent and risky. Objectives: Primary: To evaluate the effect of the implementation of the I-PASS® transfer program on the reduction in the frequency of medical attention errors in intensive pediatric therapies in the public hospitals setting. Secondary: 1) Measure the effect of the intervention in increasing the frequency of use of key elements of high quality verbal and written communication during the transfer of patients by health professionals. 2) To explore the effect of the intervention on the culture of patient safety among health professionals who assist pediatric patients in areas of clinical hospitalization. Material and Methods: Design: Staged clinical trial (Stepped Wedge) Duration: 9 months (progressive enrollment of 2 participating units every 2 months). Scope: Pediatric Intensive Care Units Subjects: health professionals involved in transfers in each institution. Intervention: Implementation of a multi-faceted evidence-based transfer package (I-PASS®) that has already been adapted for use in Argentina. The program includes multiple components, including educational training, implementation of a mnemonic verbal and written delivery rule I-PASS®, live observations of transfers to drive continuous improvement of the quality of intervention, through the feedback and a campaign of visual reinforcement materials to ensure sustainability. Events of interest: acceptance of the intervention. Frequency of preventable damages associated with medical care measured with GAPPS® as screening tools. Safety culture survey. Length of the transfer before and after the intervention.

DETAILED DESCRIPTION:
Objectives: Primary: To evaluate the effect of the implementation of the I-PASS® transfer program on the reduction in the frequency of medical attention errors in intensive pediatric therapies in the public hospitals setting. Secondary: 1) Measure the effect of the intervention in increasing the frequency of use of key elements of high quality verbal and written communication during the transfer of patients by health professionals. 2) To explore the effect of the intervention on the culture of patient safety among health professionals who assist pediatric patients in areas of clinical hospitalization. Material and Methods: Design: Staged clinical trial (Stepped Wedge) Duration: 9 months (progressive enrollment of 2 participating units every 2 months). Scope: Pediatric Intensive Care Units Subjects: health professionals involved in transfers in each institution. Intervention: Implementation of a multi-faceted evidence-based transfer package (I-PASS®) that has already been adapted for use in Argentina. The program includes multiple components, including educational training, implementation of a mnemonic verbal and written delivery rule I-PASS®, live observations of transfers to drive continuous improvement of the quality of intervention, through the feedback and a campaign of visual reinforcement materials to ensure sustainability. Events of interest: acceptance of the intervention. Frequency of preventable damages associated with medical care measured with GAPPS® as screening tools. Safety culture survey. Length of the transfer before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals (physicians only) which are currently hired as permanent staff of the participant unit
* Pediatrics medical Residents or other medical personnel in training from the pediatric ICUs enrolled.

Exclusion Criteria:

* Health professionals (physicians only) with a non permanent contract (replacements) from the pediatric ICUs enrolled.
* Health professionals other than physicians working in the participant unit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of preventable damages associated with medical care measured with GAPPS® (Global Assessment of Pediatric Patient Safety) | measured monthly along 11 months from 6/1/18 to 4/30/19
  GAPSS (retrospective chart review procedure to identify adverse events in pediatric hospitalizations) will be used to evaluate frequency of preventable adverse events in both arms

SECONDARY OUTCOMES:
IPASS usage | measured monthly along 11 months from 6/1/18 to 4/30/19
  Frequency of the use of key elements of IPASS for verbal or oral content quality of a sample of transfers (through a checklist administered by an independent observer)
Safety culture of the professionals involved in hands off: survey | At month 1 (June 2018) and at month 11 (April 2019) of data collection period.
  Safety culture survey from AHRQ will be administered to participants

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Garcia Elorrio, MD, Principal Investigator — Director. Quality and Safety in Healthcare. IECS; Luis Landry, MD, Principal Investigator — Director. Intensive Care Unit. Hospital Pedro Garrahan
Locations (5):
- Argentina (5):
  - Hospital Municipal del Niño de San Justo, San Justo, Buenos Aires
  - Hospital materno infantil héctor Quintana, San Salvador de Jujuy, Jujuy Province
  - Hospital de Niños Dr. Ricardo Gutiérrez, Buenos Aires
  - Hospital Pedro de Elizalde, Buenos Aires
  - Prof. Dr. Juan P. Garrahan, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorro-Baron F, Suarez-Anzorena I, Burgos-Pratx R, De Maio N, Penazzi M, Rodriguez AP, Rodriguez G, Velardez D, Gibbons L, Abalos S, Lardone S, Gallagher R, Olivieri J, Rodriguez R, Vassallo JC, Landry LM, Garcia-Elorrio E. Handoff improvement and adverse event reduction programme implementation in paediatric intensive care units in Argentina: a stepped-wedge trial. BMJ Qual Saf. 2021 Oct;30(10):782-791. doi: 10.1136/bmjqs-2020-012370. Epub 2021 Apr 23. PMID 33893213